CLINICAL TRIAL: NCT03056456
Title: A Study to Assess the Pharmacokinetics, Glucodynamics, Safety, and Tolerability of LY900014 in Patients With Type 1 Diabetes Mellitus on Continuous Subcutaneous Insulin Infusion Therapy
Brief Title: A Study of LY900014 Administered in Participants With Type 1 Diabetes Using an Insulin Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16727; I8B-MC-ITSC (Other: Eli Lilly and Company); 2016-004093-18 (EudraCT Number)
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): LY900014 (Treatment B) delivered via an insulin pump as a continuous infusion under the skin, with various intermittent bolus doses immediately before meals over 3-days per period.
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog) (Active Comparator): Insulin lispro (Treatment A) delivered via an insulin pump as a continuous infusion under the skin, with various intermittent bolus doses immediately before meals over 3-days per period.
  Interventions: Drug: Insulin Lispro (Humalog)

INTERVENTIONS:
Drug: LY900014 — Administered subcutaneously (SC)
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro (Humalog) — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)

SUMMARY:
This study will be conducted in participants with type 1 diabetes mellitus to investigate how the human body processes LY900014, a new blood sugar lowering insulin, and its effect on blood sugar levels when it is delivered via an insulin pump. Side effects and tolerability will be documented. The study will last about 4 to 11 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with Type 1 Diabetes Mellitus (T1DM) who are receiving insulin therapy via an approved insulin pump
* Have a screening body mass index (BMI) of greater than 18.5 to 33.0 kilograms per meter squared (kg/m²), inclusive
* Have medical and laboratory test results that are acceptable for the study
* Have had no episodes of severe hypoglycemia (requiring assistance in treatment by a second party) in the past 6 months
* Have venous access sufficient to allow for blood sampling
* Have provided written consent and are willing to follow study procedures and commit to the study duration

Exclusion Criteria:

* Are currently participating or recently participated in a clinical trial or any other type of medical research judged to be incompatible with this study
* Had blood loss of more than 500 milliliters (mL) within the last month
* Have known allergies to LY900014, insulin lispro, related compounds or any components in the study drug formulations
* Have previously participated or withdrawn from this study
* Have or used to have health problems or medical test results that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Neuss
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the time between consecutive periods, participants continued their CSII with their personal pump using Insulin lispro (Humalog) until the evening of Day -1 (after administration of the standardized dinner) of the next period when they will receive either LY900014 or Insulin lispro (Humalog), according to assigned treatment.
Pre-assignment Details: Participants were randomized to receive LY900014 and Insulin lispro (Humalog) via CSII with intermittent bolus doses, standard single-wave (SS) and standard dual-wave (SD) immediately before meals, over 3 days per period.
Groups:
- Sequence 1: Administration modes for LY900014 or Insulin lispro (Humalog) for Days 1 through 3 for breakfast (B):
  Period 1: Insulin lispro (Humalog)
  Day 1: B: SD Day 3: B: SD
  Period 2: Insulin lispro (Humalog)
  Day 1: B: SS Day 3: B: SS
  Period 3: LY900014
  Day 1: B: SD Day 3: B: SD
  Period 4: LY900014
  Day 1: B: SS Day 3: B: SS
- Sequence 2: Administration modes for LY900014 or Insulin lispro (Humalog) for Days 1 through 3 for breakfast:
  Period 1:Insulin lispro (Humalog)
  Day 1: B: SS Day 3: B: SS
  Period 2: LY900014
  Day 1: B: SS Day 3: B: SS
  Period 3: Insulin lispro (Humalog)
  Day 1: B: SD Day 3: B: SD
  Period 4: LY900014
  Day 1: B: SD Day 3: B: SD
- Sequence 3: Administration modes for LY900014 or Insulin lispro (Humalog) for Days 1 through 3 for breakfast:
  Period 1: LY900014
  Day 1: B: SD Day 3: B: SD
  Period 2: Insulin lispro (Humalog)
  Day 1: B: SD Day 3: B: SD
  Period 3: LY900014
  Day 1: B: SS Day 3: B: SS
  Period 4: Insulin lispro (Humalog)
  Day 1: B: SS Day 3: B: SS
- Sequence 4: Administration modes for LY900014 or Insulin lispro (Humalog) for Days 1 through 3 for breakfast:
  Period 1:LY900014
  Day 1: B: SS Day 3: B: SS
  Period 2: LY900014
  Day 1: B: SD Day 3: B: SD
  Period 3: Insulin lispro (Humalog)
  Day 1: B: SS Day 3: B: SS
  Period 4: Insulin lispro (Humalog)
  Day 1: B: SD Day 3: B: SD
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Received One Dose of Study Drug | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 5 (Participant deviated from 1 week maximum between consecutive periods and did not start Period 4.)
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Overall Baseline: Participants received individualized doses of LY900014 and Insulin lispro (Humalog) via CSII with various intermittent bolus doses immediately before meals, over 3 days per period.
Arm/Group | Overall Baseline
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 5 Hours(h) (AUC [0-5 h]) Following Administration of Each Study Arm With a Standard Single-wave Bolus
Description: PK: Insulin Lispro AUC(0-5h)
Time Frame: Days 1 and 3: -15, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, and 300 minutes post dose
Population: All participants who received at least one dose of both study drugs and had evaluable PK data during the breakfast test meal.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole x hour per liter (pmol*h/L)
Groups:
- LY900014 SS: Individualized doses of LY900014 delivered via CSII with intermitted bolus dose administered as standard single-wave bolus on Day 1 and 3.
- Insulin Lispro (Humalog) SS: Individualized doses of Insulin lispro (Humalog) delivered via CSII with intermittent bolus dose administered as a standard single-wave bolus on Day 1 and 3.
Arm/Group | LY900014 SS | Insulin Lispro (Humalog) SS
Number analyzed (Participants) | 24 | 24
picomole x hour per liter (pmol*h/L)
  Day 1 | 1040 (42) | 1040 (43)
  Day 3 | 1050 (47) | 1040 (48)
Statistical Analysis 1: Comparison: LY900014 SS vs Insulin Lispro (Humalog) SS; Day 1; Test type: Superiority; Ratio of Geometric LS Means = 1, 90% CI 2-sided [0.810 to 1.23]
Statistical Analysis 2: Comparison: LY900014 SS vs Insulin Lispro (Humalog) SS; Day 3; Test type: Superiority; Ratio of Geometric LS Means = 1.01, 90% CI 2-sided [0.817 to 1.25]

2. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 5 Hours (AUC [0-5 h]) of Following Administration of Each Study Arm With a Standard Dual-wave Bolus
Description: PK: Insulin Lispro AUC(0-5h)
Time Frame: as for outcome 1
Population: All participants who received both study drugs and had evaluable PK during the breakfast test meal.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Groups:
- LY900014 SD: Individualized doses of LY900014 delivered via CSII with intermitted bolus dose administered as standard dual-wave bolus on Day 1 and 3.
- Insulin Lispro (Humalog) SD: Individualized doses of Insulin lispro (Humalog) delivered via CSII with intermitted bolus dose administered as standard dual-wave bolus on Days 1 and 3.
Arm/Group | LY900014 SD | Insulin Lispro (Humalog) SD
Number analyzed (Participants) | 22 | 22
pmol*h/L
  Day 1 | 985 (48) | 956 (46)
  Day 3 | 1010 (53) | 969 (48)
Statistical Analysis 1: Comparison: LY900014 SD vs Insulin Lispro (Humalog) SD; Day 1; Test type: Superiority; Ratio of Geometric LS Means = 1.03, 90% CI 2-sided [0.808 to 1.31]
Statistical Analysis 2: Comparison: LY900014 SD vs Insulin Lispro (Humalog) SD; Test type: Superiority — Day 3; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [0.820 to 1.32]

3. Secondary Outcome: Glucodynamics (GD): Change From Baseline Area Under the Concentration Curve From Time Zero to 5 Hours (AUC [0-5h]) of Glucose Relative to Mixed Meal Tolerance Test Following Administration of Each Study Arm With a Standard Single-wave Bolus
Description: GD: Change from baseline in AUC (0-5h) of glucose relative to mixed meal tolerance test (MMTT).
Time Frame: Days 1 and 3: -30, -15, 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180,195, 210, 225, 240, and 300 minutes post dose
Population: All participants who received at least one dose of both study drugs and had evaluable GD during the breakfast test meal. Last observation carried forward (LOCF) was used for last observed glucose values prior to treatment intervention for hypoglycemic or hyperglycemic events.
Measure: Mean (Standard Deviation); unit: milligrams * hour/deciliter (mg*h/dL)
Groups:
- LY900014 SS: Individualized doses of LY900014 delivered via CSII with intermitted bolus dose administered as standard single-wave bolus on Days 1 and 3.
- Insulin Lispro (Humalog) SS: Individualized doses of Insulin lispro (Humalog) delivered via CSII with intermitted bolus dose administered as standard single-wave bolus on Days 1 and 3.
Arm/Group | LY900014 SS | Insulin Lispro (Humalog) SS
Number analyzed (Participants) | 24 | 24
milligrams * hour/deciliter (mg*h/dL)
  Day 1 | 16.8 (182) | 38.9 (186)
  Day 3 | 140 (223) | 175 (152)

4. Secondary Outcome: Glucodynamics (GD): Change From Baseline Area Under the Concentration Curve From Time Zero to 5 Hours (AUC [0-5 h]) of Glucose Relative to MMTT Following Administration of Each Study Arm With a Standard Dual-wave Bolus
Description: GD: Change from baseline in AUC (0-5h) of glucose relative to MMTT.
Time Frame: Day 1 and 3: -30, -15, 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180,195, 210, 225, 240, and 300 minutes post dose
Population: All participants who received at least one dose of both study drugs and had evaluable GD data during the breakfast test meal. LOCF was used for last observed glucose values prior to treatment intervention for hypoglycemic or hyperglycemic events.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Groups:
- LY900014 SD: Individualized doses of LY900014 delivered via CSII with intermitted bolus dose administered as standard dual-wave bolus on Days 1 and 3.
- Insulin Lispro (Humalog) SD: Individualized doses of Insulin lispro (Humalog) delivered via CSII intermitted bolus dose administered as standard dual-wave bolus on Days 1 and 3.
Arm/Group | LY900014 SD | Insulin Lispro (Humalog) SD
Number analyzed (Participants) | 22 | 22
mg*h/dL
  Day 1 | -1.87 (225) | 106 (178)
  Day 3 | 188 (234) | 286 (221)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (Up to 11 weeks)
Groups:
- LY900014: LY900014 administered via CSII
- Humalog: Humalog administered via CSII
- Open-label Humalog: Humalog administered via CSII as post-blinded study standard of care.
Arm/Group | LY900014 | Humalog | Open-label Humalog
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 19/24 | 18/24 | 10/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=24) | Humalog (N=24) | Open-label Humalog (N=24)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (6) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (2) | 2 (5)
Fatigue (General disorders) | 4 (5) | 2 (5) | 0 (0)
Hunger (General disorders) | 2 (3) | 1 (1) | 3 (6)
Headache (Nervous system disorders) | 10 (23) | 9 (15) | 5 (5)
Tremor (Nervous system disorders) | 1 (1) | 2 (3) | 3 (4)
Restlessness (Psychiatric disorders) | 6 (14) | 7 (20) | 6 (10)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Rapid-Single wave bolus data is not reported as the target fasting blood glucose was not achieved, which prevented many participants from taking part in the MMTT for Day 2 resulting in unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03056456/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03056456/SAP_001.pdf